CLINICAL TRIAL: NCT00594711
Title: Monoamine Transporter Function and Autonomic Regulation During Psychodynamic Psychotherapy
Status: Completed | Type: Observational
Sponsor: Kuopio University Hospital (Other)
Collaborators: University of Eastern Finland (Other)
Responsible Party: Principal Investigator, Taru Grohn, Pirjo Saarinen, Kuopio University Hospital
Other Study IDs: KUH5703410; 118/9/00
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Last update posted 2011-10-31 (Estimated); Status verified 2011-10

CONDITIONS: Depression
Keywords: Psychotherapy; depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA, creatine, B-vitamin,BP from blood samples.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Case-group
- 2: Control-group

SUMMARY:
Outcome of psychodynamic psychotherapy measured by [123I] nor-B-CIT SPET imaging

Background Psychodynamic psychotherapy is a widely practised form of psychotherapy in the treatment of depression. There is evidence that serotonin transporter (SERT) densities are altered in depression. Preliminary observations have suggested that SERT function may recover in connection with dynamic psychotherapy.

The objective was to determine whether SERT densities change in relation to clinical recovery during psychodynamic psychotherapy.

DETAILED DESCRIPTION:
N=26

Method Twenty six drug-naïve currently depressed (moderate/severe) patients with no previous treatment were recruited for the study. The baseline study included a group of 18 healthy controls. The patients were randomised into psychotherapy and waiting-list control groups. For controls, psychotherapy was started after a 6-month waiting period. [123I] nor-B-CIT SPET imaging was performed at baseline and after 12 months of psychotherapy. For the controls, additional imaging was performed after the 6-month waiting period.

ELIGIBILITY:
Inclusion Criteria:

* depression

Exclusion Criteria:

* antidepressive medication

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patiens of clinic
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2000-01; Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pirjo Saarinen, Ph.D., Principal Investigator — Kuopio University Hospital; Johannes Lehtonen, Ph.D, Study Director — Kuopio University Hospital; Lehto Soili, MD, Study Chair — Kuopio University Hospital; Minna Valkonen-Korhonen, Ph.D, Study Chair — Kuopio University; Pasi Ahola, MD, Study Chair — Kuopio University; Mikko Joensuu, MD, Study Chair — Kuopio University Hospital; Tommi Tolmunen, Ph.D., Study Chair — Kuopio University Hospital

REFERENCES:
- [Derived] Joensuu M, Ahola P, Knekt P, Lindfors O, Saarinen P, Tolmunen T, Valkonen-Korhonen M, Vanninen R, Jaaskelainen T, Virtala E, Kuikka J, Tiihonen J, Lehtonen J. Baseline symptom severity predicts serotonin transporter change during psychotherapy in patients with major depression. Psychiatry Clin Neurosci. 2016 Jan;70(1):34-41. doi: 10.1111/pcn.12335. Epub 2015 Sep 22. PMID 26311446